CLINICAL TRIAL: NCT01500317
Title: Comparison of the Effects of Tapentadol and Oxycodone on Gastrointestinal and Colonic Transit in Humans
Acronym: tap-oxy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 11-002334; Pharmacodynamic study (Other: Mayo Clinic); UL1RR024150 (NIH)
Record Dates: First submitted 2011-05-20; First posted 2011-12-28 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Effects of 2 Mu-opiates on Gastrointestinal Transit
Keywords: tapentadol; oxycodone; mu-opiate; stomach; small intestine; colon; motility; nausea; constipation
MeSH Terms: conditions — Nausea; Constipation | interventions — Tapentadol; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tapentadol (Active Comparator): 75 mg tapentadol tid
  Interventions: Drug: Tapentadol
- Oxycodone (Active Comparator): 5 mg oxycodone tid
  Interventions: Drug: Oxycodone
- Placebo (Placebo Comparator): Placebo tid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tapentadol — Subjects received tapentadol immediate release formulation, 75 mg three times per day (tid) for 48 hours.
  Other Names: Tapentadol brand name: Nucynta
  Arms: Tapentadol
Drug: Oxycodone — Subjects received oxycodone immediate release formulation, 5 mg three times per day (tid) for 48 hours.
  Other Names: Dazidox; ETH-Oxydose; Endocodone; Oxecta; Oxy IR; Oxycontin; Oxyfast; Percolone; Roxicodone
  Arms: Oxycodone
Drug: Placebo — Subjects received placebo three times per day (tid) for 48 hours.
  Arms: Placebo

SUMMARY:
Tapentadol is FDA approved for the treatment of moderate to severe acute pain. Due to the dual mechanism of action as an opioid agonist and norepinephrine reuptake inhibitor, there is potential for off label use in chronic pain.

Tapentadol is a new molecular entity that is structurally similar to tramadol. Tapentadol is a centrally-acting analgesic with a dual mode of action as an agonist at the mu-opioid receptor and as a norepinephrine reuptake inhibitor. These two actions are synergistic in pain relief. While its action reflects aspects of tramadol and morphine, its ability to control pain is more on the order of hydrocodone and oxycodone.

Its dual mode of action provides analgesia at similar levels of more potent narcotic analgesics such as hydrocodone, oxycodone, and meperidine with a more tolerable side effect profile. Clinical studies showed that tapentadol effectively relieves moderate to severe pain in various pain care settings. In addition, it was reported to be associated with significantly fewer treatment discontinuations due to a significantly lower incidence of gastrointestinal-related adverse events compared with equivalent doses of oxycodone. The combination of these reduced treatment discontinuation rates and tapentadol efficacy for the relief of moderate to severe nociceptive and neuropathic pain may offer an improvement in pain therapy by increasing patient compliance with their treatment regimen.

DETAILED DESCRIPTION:
Single center, parallel group, randomized controlled trial of tapentadol, oxycodone and placebo effects on gastrointestinal and colonic transit in healthy human volunteers

ELIGIBILITY:
Healthy volunteers Inclusion criteria

1. Males and non-pregnant, non-breastfeeding females
2. 18-65 years old

Exclusion criteria

1. Use of any mu-opioid agent in the last 3 months
2. Structural or metabolic diseases/conditions that affect the gastrointestinal system, or functional gastrointestinal disorders. For screening the shortened screening version of the Bowel Disease Questionnaire (Appendix) will be used to exclude subjects with dyspepsia, irritable bowel syndrome or significant gastrointestinal symptoms. Of 19 questions, participants have to have three or less positives to be eligible to participate.
3. Unable to withdraw medications 48 hours prior to the study :

   * Alter GI transit including laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, tricyclic antidepressants, selective serotonin re-uptake inhibitors (SSRIs) and newer antidepressants.
   * Analgesic drugs including opiates, nonsteroidal anti-inflammatory drugs (NSAIDs), COX 2 inhibitors
   * SSRI NOTE: Low stable doses of thyroid replacement, estrogen replacement, low dose aspirin for cardioprotection and birth control pills or depot injections are permissible.
4. Female subjects who are pregnant or breast feeding.
5. Clinical evidence (including physical exam, ECG, hemoglobin level and review of the medical history) of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric, or other disease that interfere with the objectives of the study.
6. Subjects who are considered by the investigator to be alcoholics not in remission or known substance abusers.
7. Subjects who have participated in another clinical study within the past 30 days
8. History of porphyria, renal (creatinine > 1.5mg/dL) or significant liver impairment (transaminases, alkaline phosphatase of gamma-glutamyl transpeptidase (GGT) >2 times upper limit of normal)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tapentadol | Oxycodone | Placebo
Started | 13 | 12 | 13
Completed | 10 | 10 | 13
Not Completed | 3 | 2 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol | Oxycodone | Placebo | Total
Number analyzed (Participants) | 13 | 12 | 13 | 38
Age Continuous [Mean (Standard Deviation); unit: years] | 34.99 (7.82) | 33.26 (12.94) | 39.48 (12) | 35.98 (11.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 10 | 28
  Male | 4 | 3 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 13 | 38
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.27 (4.88) | 27.36 (6.11) | 25.16 (4.88) | 26.23 (5.23)

OUTCOME MEASURES:

1. Primary Outcome: Colonic Transit, Geometric Center at 24 Hours
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 12 | 13
units on a scale | 2.06 (0.67) | 2.07 (0.6) | 2.17 (0.739)

2. Secondary Outcome: Colonic Geometric Center at 8 and 48 Hours
Description: as for outcome 1
Time Frame: 8 hours, 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tapentadol | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 12 | 13
units on a scale
  Colonic geometric center at 8 hr | 0.78 (0.589) | 0.75 (0.54) | 0.79 (0.98)
  Colonic geometric center at 48 hr | 3.59 (1.16) | 3.51 (0.82) | 3.742 (0.83)

3. Primary Outcome: Gastric Emptying Half-time (t1/2) at 24 Hours
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tapentadol | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 12 | 13
minutes | 159.2 (46.45) | 155.2 (38.44) | 124.7 (39.08)

4. Secondary Outcome: Colonic Filling at 6 Hours
Description: Percent of the radio-labeled meal that reached the colon at 6 hours, indirectly reflecting small bowel transit time.
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: percentage of radio-labeled meal
Arm/Group | Tapentadol | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 12 | 13
percentage of radio-labeled meal | 35.55 (32.3) | 38.6 (19.5) | 65.54 (26.1)

5. Secondary Outcome: Ascending Colon Emptying (AC t1/2)
Description: Ascending colon emptying t1/2 will be estimated by power exponential analysis of the proportionate emptying over time of counts from the colon. The primary data for this analysis will be the proportion of decay and depth-corrected counts in the ascending colon on the hourly scans on the first day of transit measurement and the 24 hour data.
Time Frame: Over the first 24 hours after ingestion of the radioisotopically labeled charcoal particles
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tapentadol | Oxycodone | Placebo
Number analyzed (Participants) | 13 | 12 | 13
hours | 21.92 (9.89) | 19.3 (6.27) | 17.88 (6.21)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during visits, and participants were contacted 5-7 days following the last dose of study medication to determine if any adverse events had occurred.
Arm/Group | Tapentadol | Oxycodone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 10/13 | 4/12 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tapentadol (N=13) | Oxycodone (N=12) | Placebo (N=13)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Light-headed (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No